CLINICAL TRIAL: NCT07258238
Title: Romanian Validation and Cross-cultural Adaptation of the QoR-15 Post-anesthetic Recovery Quality Questionnaire: The QoR-15Ro
Brief Title: Romanian Validation and Cross-cultural Adaptation of the QoR-15Ro
Acronym: QoR-15Ro
Status: Not yet recruiting | Type: Observational
Sponsor: SUUMC Central Military Hospital Dr Carol Davila (Other)
Responsible Party: Principal Investigator, Blajut Cristian, Consultant Surgeon, SUUMC Central Military Hospital Dr Carol Davila
Other Study IDs: QoR-15Ro
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Humans; Anesthesia; Recovery; Postoperative Care; Postoperative Period
Keywords: Quality of Recovery; Postoperative Recovery; QoR-15

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Optimal postoperative recovery after any surgical procedure requiring anesthesia is essential to achieving high-quality care. The Quality of Recovery questionnaire (QoR-15) was validated by its authors in 2013 in the study "Development and psychometric evaluation of a postoperative quality of recovery score: the QoR-15." This instrument enables a comprehensive evaluation by integrating traditional physiological measures with the patient's subjective perception of their health status. With the consent of the original author, the present study aims to validate the Romanian version of the questionnaire and adapt it to our clinical environment.

DETAILED DESCRIPTION:
The goal of this observational study is to validate the Romanian translation of the Quality of Recovery questionnaire (QoR-15) in adult patients undergoing surgery with anesthesia. The study aims to determine whether the Romanian version of the QoR-15 accurately measures postoperative recovery by reflecting both physical and emotional aspects of the patient's health.

The main questions it aims to answer are: Is the Romanian QoR-15 a reliable and consistent tool for evaluating postoperative recovery? AND Does the Romanian QoR-15 accurately capture the patient's own perception of their recovery after anesthesia and surgery? Participants will complete the Romanian version of the QoR-15 within the postoperative period and provide basic demographic and clinical information relevant to their recovery.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old.
* Comprehensive and sign informed consent.
* Knows and understands the Romanian language.
* Undergo a scheduled surgical intervention under any type of anesthetic procedure from the specialties of general surgery, urology, neurosurgery, plastic and reconstructive surgery.
* Score > 26 points in the Mini Mental State Examination (MMSE) test.

Exclusion Criteria:

* Patients under 18 years old.
* Not having signed the informed consent.
* Not knowing or understanding the Romanian language.
* Surgical intervention from other specialties than general surgery, urology, neurosurgery, plastic and reconstructive surgery.
* Score < 27 points in the Mini Mental State Examination (MMSE) test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our study population will consist of adult patients undergoing therapeutic or diagnostic surgical procedures in the specialties of general surgery, urology, neurosurgery, and plastic and reconstructive surgery that require anesthesia. All participants will be treated at the Central Military University Emergency Hospital "Dr. Carol Davila" in Bucharest and are expected to be transferred to the post-anesthetic recovery unit immediately after the procedure, prior to hospital discharge.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Romanian version of the Quality of Recovery 15 questionnaire: The QoR-15Ro. | 6 months
  The aim of this study is to carry out cross-cultural adaptation and validate the postoperative questionnaire QoR-15 in the Romanian environment and evaluate its validity and reliability.
  This questionnaire consists of 15 items with a total score of 150 points, where 150 points is better than 0 points for the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- The Central Military University Emergency Hospital "Dr. Carol Davila" in Bucharest, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Demumieux F, Ludes PO, Diemunsch P, Bennett-Guerrero E, Lujic M, Lefebvre F, Noll E. Validation of the translated Quality of Recovery-15 questionnaire in a French-speaking population. Br J Anaesth. 2020 Jun;124(6):761-767. doi: 10.1016/j.bja.2020.03.011. Epub 2020 Apr 15. PMID 32303379
- [Background] Morales-Ariza V, Loaiza-Aldean Y, de Miguel M, Pena-Navarro M, Martinez-Silva O, Gonzalez-Tallada A, Manrique-Munoz S, de Nadal M. Validation and cross-cultural adaptation of the postoperative quality of recovery 15 (QoR-15) questionnaire for Spanish-speaking patients: A prospective cohort study. Am J Surg. 2023 Apr;225(4):740-747. doi: 10.1016/j.amjsurg.2022.11.009. Epub 2022 Nov 17. PMID 36414472
- [Background] Kleif J, Waage J, Christensen KB, Gogenur I. Systematic review of the QoR-15 score, a patient- reported outcome measure measuring quality of recovery after surgery and anaesthesia. Br J Anaesth. 2018 Jan;120(1):28-36. doi: 10.1016/j.bja.2017.11.013. Epub 2017 Nov 22. PMID 29397134
- [Background] Myles PS, Shulman MA, Reilly J, Kasza J, Romero L. Measurement of quality of recovery after surgery using the 15-item quality of recovery scale: a systematic review and meta-analysis. Br J Anaesth. 2022 Jun;128(6):1029-1039. doi: 10.1016/j.bja.2022.03.009. Epub 2022 Apr 14. PMID 35430086
- [Background] Stark PA, Myles PS, Burke JA. Development and psychometric evaluation of a postoperative quality of recovery score: the QoR-15. Anesthesiology. 2013 Jun;118(6):1332-40. doi: 10.1097/ALN.0b013e318289b84b. PMID 23411725